CLINICAL TRIAL: NCT05694858
Title: Transdermal Microneedle Lignocaine Delivery Versus EMLA Patch for Topical Analgesia Before Venepuncture Procedure To Adults in Clinical Setting
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UKM/PPI/111/8/JEP-2022-736; FF-2022-401 (Other Grant/Funding Number: Faculty of Medicine, Universiti Kebangsaan Malaysia (UKM), Malaysia); MOSTI.D (S) 600-4/19/15 (Other Grant/Funding Number: Ministry of Science, Technology and Innovation (MOSTI), Malaysia)
Record Dates: First submitted 2023-01-10; First posted 2023-01-23 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Glaucoma; Cataract; Ophthalmological Disorder
Keywords: Microneedle; Maltose Microneedle; EMLA; EMLA-impregnated microneedle; Cataract; Glaucoma; Venepuncture
MeSH Terms: conditions — Glaucoma; Cataract; Eye Diseases | interventions — Lidocaine, Prilocaine Drug Combination; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lignocaine-Embedded Microneedle Patch (Experimental): A biodegradable maltose microarray needle (MAN) patch loaded with 12.5 mg lignocaine will be applied on the dorsum of the participant's hand for 30 minutes. Venepuncture will be carried out after 30 minutes.
  Interventions: Combination Product: Lignocaine-loaded maltose microneedle array patch
- EMLA 5% Patch (Active Comparator): 1 finger-tip unit (FTU) of EMLA containing 12.5 mg lignocaine and 12.5 mg prilocaine will be applied on the dorsum aspect of the participant's hand. This will then be covered by a Polyvinyl Alcohol (PVA)-Polyethylene Terephthalate (PET) adhesive and left in place for 30 minutes. Venepuncture will be carried out after 30 minutes.
  Interventions: Drug: EMLA 5% patch

INTERVENTIONS:
Combination Product: Lignocaine-loaded maltose microneedle array patch — A biodegradable maltose microneedle array patch containing 12.5 mg lignocaine that will be applied on the participant's dorsal aspect of the hand for 30 minutes prior to venepuncture.
  Other Names: Lignocaine-embedded microneedle array patch
  Arms: Lignocaine-Embedded Microneedle Patch
Drug: EMLA 5% patch — EMLA 5% cream applied on the dorsum of the participant's hand which will be subsequently covered with PVA-PET adhesive for 30 minutes prior to venepuncture
  Other Names: Standard EMLA 5% patch
  Arms: EMLA 5% Patch

SUMMARY:
Microneedle (MN) is a mimic of a hypodermic needle, composed of hundreds of micron-sized, out-of-plane protrusions, typically arranged in arrays on a patch that can be applied onto the skin. MN can be fabricated from a variety of materials, preferably biocompatible polymers. Maltose, a natural carbohydrate, is a safe and biocompatible product that can be fabricated into MNs that are biodegradable and soluble within several minutes. Besides, local anaesthetic agents such as lignocaine can be impregnated within the MN matrix, facilitating its transdermal delivery more efficiently which results in enhanced efficacy. So far, maltose MN efficacy in enhancing the transdermal drug delivery (TDD) of lignocaine and thus reducing the pain experienced by healthy patients requiring venepuncture prior to routine eye surgeries (phacoemulsification, trabeculectomy etc) has not been extensively studied. Hence, the objectives of this research are: 1) To evaluate the safety profile of lignocaine-embedded microneedle patch as a means of pain reduction in adult patients requiring routine vein-puncturing procedures; 2) To assess the pharmacokinetic (PK) parameters of lignocaine in the systemic circulation when the transdermal lignocaine delivery is enhanced through microneedle usage; 3) To compare the efficacy of lignocaine-embedded microneedle patch with standard 5% Eutectic Mixture of Local Anesthetics (EMLA) dermal patch for pain reduction during venepuncture procedure based on mean changes in VAS scores and skin algesimeter index (pharmacodynamic (PD) study).

DETAILED DESCRIPTION:
This is a prospective, phase I/II, randomized, triple-blind (participants and care providers), two-parallel group, active controlled trial.

This study is divided into two phases:

A) Phase I: Non-randomized single-centre open-label single group clinical trial to primarily assess the safety and tolerability of lignocaine-impregnated microneedle in adult patients undergoing routine vein-puncturing related procedures (pharmacokinetic (PK) study).

B) Phase II: A randomized single centre double blind two parallel group active controlled clinical trial to assess the efficacy of lignocaine-impregnated microneedle compared to 5% EMLA dermal patch (Pharmacodynamic (PD) study).

I) Phase I Study

For phase I of the research, the safety and tolerability of 12.5mg lignocaine-embedded microneedle on a small number of adult patients (20 patients; 10 males and 10 females) without hepatic or renal dysfunction will be assessed.All participants of this phase I will be healthy patients who undergo cataract or glaucoma surgeries who will be recruited from the Hospital Canselor Tuanku Muhriz (HCTM), Universiti Kebangsaan Malaysia (UKM) ophthalmology outpatient clinic. Pre-treatment fasting is not required for all participants.

On the day of the study, each potential participant will be screened for study eligibility based on our pre-specified inclusion and exclusion criteria. An interim abridged medical history will be taken from each participant and their list of medications will be reviewed. Vital signs (systolic and diastolic blood pressures, oral temperature, pulse and respiratory rates) will be taken and targeted clinical examinations will be performed by the medical officers to assess the overall health of the participants.

After the 12.5mg lignocaine-impregnated microneedles have been applied to the designated sites, intravenous cannula will be placed on the dorsal aspect of the participant's right hand. Approximately 3.0 ml venous blood samples will then be withdrawn from the antecubital fossa at each t=0, 30, 60, 90, 120, 180 minutes and collected into separate 3.5-ml of plastic blood collection tube with accelerator & separator gel (BD™, New Jersey, USA). Heparinized saline will be periodically infused to ensure that the cannula lumen remains patent throughout the sampling periods. The blood samples will then be sent to the Malaysian Institute of Chemistry for lignocaine concentration measurements using the validated Gas Chromatography Nitrogen Phosphorus Detector (GC-NPD) methodology.

The participants will be allowed to return home after the last blood sample is taken at t=180. The participants will be further monitored for any adverse events (AEs) such as redness, pain, itchiness, blistering, etc (local reactions) and light-headedness, euphoria, tinnitus, diplopia etc. (systemic reactions), serious adverse events (SAEs) and suspected unexpected serious adverse reactions (SUSARs) for up to 48 hours via telephone calls.

The pharmacokinetic data will be first summarized in mean / standard deviation or median / interquartile range for continuous data and count and percentage for categorical data. The pharmacokinetic parameters (Area under the curve until time = infinity (AUCinf), Area under the curve until time t (AUCt), Cmax, Cmin, tmax, t1/2, volume of distribution (Vd), Clearance (Cl)) of lignocaine will be evaluated using blood samples obtained at times t=0, 30, 60, 90, 120, and 180 minutes after the application of lignocaine-impregnated MN patch. The intraindividual and interindividual variations of the pharmacokinetic parameters will be evaluated using coefficient of variation (CV) and these will be classified as low (CV≤10%), moderate (CV ≈ 25%) and high (CV>40%).63 The pharmacokinetic data will be analysed using the non-linear mixed effect models based on two-compartmental model which will be implemented on NONMEM® version VI (Icon Development Solutions, Ellicott City, Maryland, USA). The influence of clinically relevant covariates such as participant's age, gender, BMI and others on pharmacokinetic parameters will be evaluated in a stepwise fashion. First-order conditional likelihood (FOCE INTER on NONMEM) will be used to fit the data and model selection will be dependent upon the likelihood ratio test, the estimates of pharmacokinetic parameters and their 95% confidence intervals and goodness-of fit measures.

II) Phase II Study

For phase II of the research lidocaine-impregnated microneedle patch will be used as the experimental agent under study (i.e. studied agent). As a comparator, the standard EMLA patch which is a eutectic emulsion mixture of lidocaine and prilocaine at 1:1 ratio (i.e. each gram of EMLA cream contains lidocaine and prilocaine, 25 mg each). A eutectic mixture has a lower melting temperature than each constituent's melting temperature. The anaesthetic efficacy of EMLA cream will be assessed via pain induced by venipuncture and the primary endpoint are the participant's VAS score and skin algesimeter index measured 30 minutes after either lignocaine-impregnated patch or EMLA patch application.

1. Randomization Procedure and Blinding (Masking) of Trial Participants

   For random allocation, block randomization procedure with varying block size (permuted block) will be utilized to guarantee that both intervention groups will have an equal number of trial participants. This will be carried out by the trial statistician using the R package, blockrand version 1.50 which will be implemented on R platform. The list of generated random numbers will be used to allocate the study participants to either intervention or control branch. The allocation sequence generated will be kept in a password-protected document that is only accessible to the statistician to maintain allocation concealment. To further ensure the adequacy of allocation concealment, randomisation code will not be revealed until the potential trial participants have been definitively enrolled into the trial, which will be after all baseline measurements are made and all eligibility criteria are deemed fulfilled by the study recruiters. In addition, allocation concealment is further safeguarded by ensuring identity of the allotted treatment is only revealed to the interventionist (i.e. the person who will be administering the intervention) via secured telephone calls (central randomization). Consecutive recruitments will be made until the final intended sample size is achieved.

   For this study, the outcome assessors and care providers (may be the same individual) will be masked to the identity of interventions (single blinding / single masking). Only the statistician and interventionist/procedurist will be unmasked to the study interventions. Furthermore, unique ID code to indicate each treatment sequence assignment will be generated and utilised to ensure that the unintentional / intentional unmasking of one trial participant will not compromise the integrity of blinding for the rest of study participants. The primary unblinded trial persons (subjects, the statistician and the procedurist/interventionist) are instructed not to divulge the identity of the allotted treatments to other blinded trial personnel. The success of blinding will be determined by asking the blinded trial persons to guess the identity of interventions received and then compare the results obtained with what would be anticipated by chance. Blinding indices such as James' Blinding Index or Bang's blinding Index could also be calculated to objectively assess whether blinding has been successfully achieved in this trial.
2. Administration of Lignocaine-embedded Microneedle (intervention) and EMLA (control) patches

   Prior to the administration of intervention/control, relevant clinic-demographic profiles (age, gender, ethnicity, anthropometric measurements, presence of comorbidities, the types of eye surgeries received etc.) will be recorded and entered in the case report forms (CRFs) that are specifically designed for this study. This research study uses lignocaine embedded microneedles. The comparison of pharmacodynamic properties (i.e. efficacy) between 12.5 mg lignocaine delivered through direct embedment within the microneedle matrix and standard 5% EMLA dermal patch containing 1 finger-tip- unit (FTU=0.5g) of 12.5mg lignocaine and 12.5mg prilocaine will be assessed via VAS score and skin algesimeter index for the pain induced by venepuncture.

   The window period given to lignocaine for it to be effective will be based on the usual clinical practice observation where it is usually applied for 30 minutes prior to venepuncture. The rationale behind it is due to logistical issues and for the day care's operational convenience. Nevertheless, in a busy clinical setting, the application time is sometimes shortened to 15 minutes for a slight anaesthetic effect. Thus, we postulate that, with the aid of microneedle, the time to onset of action for lignocaine could be greatly reduced resulting in a much more reduced pain sensation when the clinical assessment is carried out 30 minutes after treatment application.

   The administrator of interventions (procedurist) will identify and draw a grid of 1cm × 1cm at the dorsum hand, which will serve as an ideal site for venepuncture. The procedurist will then apply the lignocaine-impregnated microneedle patch. After a 30-minute application time, the attending medical officer will perform venepuncture line using a 21-gauge (G) hypodermic needle inserted into the vein in the dorsal aspect of the participant's hand.

   For the participants allotted to the standard 5% EMLA dermal patch, 1 FTU of 5% EMLA cream will be applied and covered with a piece of adhesive to form a dermal patch. This will be applied for 30 minutes on the dorsum of the hand which will be cleaned and dried first. This application is equivalent to 12.5mg lignocaine and 12.5mg prilocaine. The EMLA patch will be firmly applied to the designated area (dorsal aspect of the hand).

   During the trial day, the participants will not be allowed to take any analgesic medications (NSAID, Opioids, Paracetamol) since they will modulate the level of pain experienced by the participants due to the received interventions. Other medications and concomitant care will be permitted during the trial.
3. Pain Assessment

The study participants will first be guided on the operating manual for a 10-points, 100mm VAS pain score by an outcome assessor. The participants will be presented with a ruler that contains 100-mm slots with "No Pain" written on the left side and "Worst Pain" on the opposite right side. The study participants will then be asked to move and place the slider in the slot that accurately describes his/her pain at the following time points: 1) within 5 minutes after application of lignocaine-impregnated MN patch and before venepuncture (baseline VAS score); 2) within 5 minutes after venepuncture. The investigator/outcome assessor, who is blinded to the subject intervention arm will record the location of the slot where the slider is placed in millimetres (mm), clearly printed on the ruler's reverse side and this will be the participant's VAS score. Throughout the process, there will be a trained investigator standing by to assist the verification of the pain scale and to aid the participants who require additional assistance.

For a subset of randomly selected patients, before applying MN patch and EMLA Cream, the patients will be attached with the PainMonitor™ (Med-Storm Innovation AS, Oslo, Norway) device whereby the electrodes will be attached to the hypothenar eminence of the opposite hand not receiving venepuncture. The procedurist will set up this machine and application before the interventions are commenced. The skin conductance peaks (in microSiemens (μS) and the skin algesimeter index (in microSiemens per second (μS/s)) will be recorded by the outcome assessor who will be blinded to the subject intervention arm. Those parameters indicate the skin's sympathetic nerve block induced by the topical anaesthetic. The measurement time points start from the point of intervention and the recordings continued for at least 15 seconds.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old and above
* Patients requiring venepuncture for blood investigations before ophthalmological procedures

Exclusion Criteria:

* Patient with a previous history of sensitization or allergy to lignocaine.
* Patient with a previous history of allergy to materials used in the study i.e., plaster, electrodes, maltose, Polyvinyl Alcohol (PVA), and Polyethylene Terephthalate (PET)
* Patient exposed to analgesic usage within 24 hours prior to the procedure
* Generalized skin disorder/ rash
* Agitated/ fretful / uncooperative patient
* Uncommunicative/deaf/mute patients
* Patients on hypnotics, or chronic pain relief medications
* Patients with psychiatric conditions
* Patients with hepatic impairment
* Patients who are on CYP450 3A4, 3A5 or 1A2-inducing or inhibiting drugs (erythromycin, ciprofloxacin, amiodarone etc.) or pharmacotherapeutic agents that affect hepatic blood flow (metoprolol) since both may affect the metabolism of lignocaine
* Failed first/single attempt at venepuncture after the application of the LEMAP or PET patch for control arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Score (VAS) | The measurements will be made at 1 minute after venepuncture which will be inserted following EMLA-impregnated microneedle patch or standard EMLA patch application]
  VAS score is measured in a continuous scale (range 0-100). It is obtained using a Med-05-100 VAS Pain Scale ruler (Schlenker Enterprises Ltd, Lombard, USA) with 0-100 mm slider. It is measured based on the pain experienced on the venepunctured hand. Higher VAS score indicates greater intensity or degree of pain whilst lower VAS score indicates lesser pain intensity.
Skin Conductance Algesimeter Index | The measurements will be made at 1 minute after venepuncture which will be inserted following EMLA-impregnated microneedle patch or standard EMLA patch application]
  The skin conductance peaks per second, measured in microSiemens per second (μS/s), is obtained using PainMonitor™ (Med-Storm Innovation AS, Oslo, Norway) device on the hypothenar eminence of the opposite hand not receiving venepuncture. Higher skin conductance algesimeter index indicates greater pain intensity and lower values indicate lesser pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: FOOK CHOE CHEAH, MD, PhD, MRCPCH, Principal Investigator — FACULTY OF MEDICINE, UNIVERSITI KEBANGSAAN MALAYSIA (UKM); AZRUL AZLAN BIN HAMZAH, BSc, PhD, Principal Investigator — INSTITUTE OF MICROENGINEERING AND NANOELECTRONICS, UNIVERSITI KEBANGSAAN MALAYSIA
Locations (1):
- Hospital Canselor Tuanku Muhriz, Universiti Kebangsaan Malaysia (Ukm Medical Centre), Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized and de-identified participants' clinical and trial outcome data will be shared through the Harvard Dataverse Repository (https://dataverse.harvard.edu/). The full statistical codes used for trial data cleaning, transformation and analysis will be made available on the GitHub repository.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The study protocol, including a statistical analysis plan, will be published in full in an open-access journal, starting after the acceptance of the protocol manuscript (tentatively by October 2025). The individual patient data will be shared after the completion of both trial phases (12th December 2026) until 11th December 2036, for a total period of 10 years.
Access Criteria: All interested readers will have access to the IPD and supporting information

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Amended Study Protocol (Version 3) (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT05694858/Prot_SAP_ICF_000.pdf
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Amended Trial Protocol (Version 3.0) (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT05694858/Prot_SAP_ICF_001.pdf